CLINICAL TRIAL: NCT01261650
Title: Influence of Transcranial Direct Current Stimulation of the Primary Motor Cortex on Pain Sensation in Patients Suffering From Fibromyalgia Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There could not be enough patients recruited
Sponsor: Karl Landsteiner Institute of Remobilization and Functional Health (Other)
Responsible Party: Karl Landsteiner Institute of Remobilization and Functional Health, Institute of Physical Medicine and Rehabilitation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FIBRO 1
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Fibromyalgia
Keywords: widespread chronic pain, transcranial direct current stimulation, fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcranial direct current stimulation (Active Comparator): transcranial direct current stimulation of the primary motor cortex
  Interventions: Device: transcranial direct current stimulation
- sham treatment (Sham Comparator)
  Interventions: Device: sham treatment

INTERVENTIONS:
Device: transcranial direct current stimulation
  Arms: transcranial direct current stimulation
Device: sham treatment
  Arms: sham treatment

SUMMARY:
Fibromyalgia is a common chronic pain syndrome characterized by bad treatable chronic widespread pain present at a similar level for at least 3 months. The aim of this study is to examine if 3 weeks of transcranial direct current stimulation is a suitable therapy to reduce chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an established diagnosis of fibromyalgia according to the 1990 criteria of the "American College of Rheumatology"
* Symptoms have been present at a similar level for at least 3 months
* Stable medication for at least 2 months
* visual analog scale ≥ 3 (0=no pain; 10=worst possible pain)
* The patient does not have a disorder that would otherwise explain the pain

Exclusion Criteria:

* Alcohol/substance abuse
* Pregnancy
* Neuropsychiatric disorders
* Metal implants near stimulation area
* Cardiac pace maker
* Local injuries
* Inflammatory rheumatic disease
* Acute tumor
* Acute fracture
* Well-defined neuropathic induced pain

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12

PRIMARY OUTCOMES:
Visual Analoge Scale | Difference Baseline - after treatment

SECONDARY OUTCOMES:
Quality of Life - SF-36 | baseline / after treatment / 1 , 2, 3 months after treatment
Fibromyalgia Impact Questionaire | baseline / after treatment / 1,2,3, months after treatment
IL-10 ELISA | baseline / after treatment / 1,2,3, months after treatment
Visual analog scale | 1,2,3 months after treatment
IL-6 ELISA | baseline / after treatment / 1,2,3, months after treatment
IL-4 ELISA | baseline / after treatment / 1,2,3, months after treatment
TNF-alpha ELISA | baseline / after treatment / 1,2,3, months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quittan, PhD, Principal Investigator — Karl Landsteiner Institute of Remobilisation and functional Health
Locations (1):
- Karl Landsteiner Institute of Remobilisation and Functional Health, Vienna, Vienna, Austria